## **Cover Page**

## Study title

The Effects of Low-Volume High Intensity Interval Training and Circuit Training on Maximal Oxygen Uptake

Trial Number: NCT03700671

**Date:** 11/05/17

Health

&



## Study title

| The Effects of | Low-Volume High | Intensity Interval | Training and | Circuit Train | ing on Maxima | l Oxyger |
|---|---|---|---|---|---|---|
| Uptake | | | | | | |

| | take |
|---|---|
| Tri | al Number: NCT03700671 |
| Da | te: 11/05/17 |
| | Informed Consent Form |
| ı | Name of test(s) |
| | The participant should complete this sheet himself / herself |
| 1. | Have you completed the pre-exercise medical questionnaire? YES / NO |
| 2. | Do you understand that your information will be treated as confidential? YES / NO |
| 3. | Have you read the participant information sheet? YES / NO |
| 4. | Have you had the opportunity to ask questions and discuss the test? YES / NO |
| 5. | Have you received satisfactory answers to all of your questions? YES / NO |
| 6. | Have you received adequate information about the test? YES / NO |
| | With whom have you discussed the nature of the test? |
| | Do you understand that you may withdraw from the test: • At any time • Without needing to give reason • Without prejudice YES / NO |
| 9. | I have read, discussed and fully understand the requirements, procedures, and potential risks involved in the test and give consent for my participation. |
| Si | ignature Date |
| Те | est Administrator Date |
| Pa | rent/Guardian if Minor |